CLINICAL TRIAL: NCT00074321
Title: A Phase I And Pharmacogenetic Study Of CPT-11, Oxaliplatin, And Capecitabine In Patients With Solid Tumors
Brief Title: Irinotecan, Oxaliplatin, and Capecitabine in Treating Patients With Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01444; MC0311; NCI-6240; CDR0000344367; MAYO-MC0311
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Irinotecan; Oxaliplatin; Capecitabine

ARMS (1):
- Arm I (Experimental): Patients receive irinotecan hydrochloride IV over 90 minutes and oxaliplatin IV over 2 hours on day 1 and capecitabine PO QD on days 2-15. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: irinotecan hydrochloride; Drug: oxaliplatin; Drug: capecitabine; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: capecitabine — Given PO
  Other Names: CAPE; Ro 09-1978/000; Xeloda
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Drugs used in chemotherapy, such as irinotecan, oxaliplatin, and capecitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug may kill more tumor cells. This phase I trial is studying the side effects and best dose of irinotecan, oxaliplatin, and capecitabine in treating patients with unresectable solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To define the maximally tolerated dose of the combination of CPT-11 (irinotecan hydrochloride), oxaliplatin, and capecitabine in three different populations, based on UDP glucuronosyltransferase 1 family, polypeptide A1 (UGT1A1) genotype (6/6, 6/7, and 7/7).

II. To identify any activity of this treatment combination in patients with metastatic cancer.

III. To examine the differences in the toxicity profile, especially pertaining to hematologic and gastrointestinal (GI), and the maximally tolerated dose of the combination of CPT-11, oxaliplatin and capecitabine with respect to the UGT1A1 haplotypes.

IV. Examine the effect of the UGT1A1 genotype on the pharmacokinetics of CPT-11 and its metabolites.

OUTLINE: This is a dose-escalation study. Patients are stratified according to UGT1A1 genotype (6/6 vs 6/7 [closed to accrual as of 8/24/06] vs 7/7).

Patients receive irinotecan hydrochloride intravenously (IV) over 90 minutes and oxaliplatin IV over 2 hours on day 1 and capecitabine orally (PO) twice daily (QD) on days 2-15. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of irinotecan hydrochloride, oxaliplatin, and capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional 6-10 patients (for a total of 12 patients) receive treatment at that dose.

After completion of study treatment, patients are followed up at 3 months.

PROJECTED ACCRUAL: A total of 54-84 patients (12-22 for stratum I, 18-28 for stratum II [closed to accrual as of 8/24/06], and 24-34 for stratum III) will be accrued for this study within approximately 4.4 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor for which there is no known standard therapy that is potentially curative or capable of extending life expectancy

  * Unresectable disease
* Willing to provide biologic specimens to determine UGT1A1 genotype
* No CNS metastases

  * Prior CNS metastases allowed provided patient was treated with surgery and/or radiotherapy and is stable for more than 8 weeks
* Performance status - ECOG 0-2
* At least 12 weeks
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL
* Bilirubin no greater than upper limit of normal (ULN) for patients with 6/6 UGT1A1 genotype (1.5 times ULN for patients with 6/7 [closed to accrual as of 8/24/06] or 7/7 UGT1A1 genotype)
* AST no greater than 3 times ULN (5 times ULN if there is liver involvement)
* Creatinine no greater than 1.5 times ULN
* No New York Heart Association class III or IV heart disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergy to platinum compounds, irinotecan, or to antiemetics or antidiarrheals appropriate for administration with study therapy
* No uncontrolled infection
* No seizure disorder
* No peripheral neuropathy grade 2 or greater
* More than 4 weeks since prior biologic therapy
* More than 4 weeks since prior immunotherapy
* No concurrent immunotherapy
* No concurrent prophylactic colony-stimulating factor therapy
* More than 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered
* No other concurrent chemotherapy
* See Disease Characteristics
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to more than 25% of the bone marrow
* No concurrent radiotherapy
* See Disease Characteristics
* No other concurrent investigational therapy
* No concurrent sorivudine, brivudine, lamivudine, or stavudine
* No concurrent enrollment in any other study involving a pharmacologic agent for symptom control or therapeutic intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2003-11; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
MTD defined as one dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients) assessed using NCI CTCAE v3.0 | 3 weeks

SECONDARY OUTCOMES:
Incidence of UTG1A1*28 polymorphism | Up to 3 months
  The overall incidence of UTG1A1*28 polymorphism will be estimated and summarized in this patient population. In addition, the incidence of this polymorphism will be explored in relation to tumor type.
Adverse events profile assessed using NCI CTCAE v3.0 | Up to 3 months
  The number and severity of all adverse events (overall, by dose level, and by tumor group) will be tabulated and summarized for the three patient groups. The grade 3+ adverse events will also be described and summarized in a similar fashion.
Toxicity profile assessed using NCI CTCAE v3.0 | Up to 3 months
  Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized in each of the two groups. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Response profile using RECIST criteria | Up to 3 months
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as table and progressive disease in the two patient populations (overall and by tumor group).
Time until any treatment related toxicity | Up to 3 months
  Will be summarized descriptively.
Time until treatment related grade 3+ toxicity | Up to 3 months
  Will be summarized descriptively.
Time until hematologic nadirs (WBC, ANC, platelets) | Up to 3 months
  Will be summarized descriptively.
Time to progression | Up to 3 months
  Will be summarized descriptively.
Time to treatment failure | From registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by the patient, assessed up to 3 months
  Will be summarized descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Goetz, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States